CLINICAL TRIAL: NCT03705000
Title: Safety and Efficacy of the Slit Stent II Lacrimal Stent for the Treatment of Nasolacrimal Duct Obstruction
Brief Title: SLlt Stent II Lacrimal Stent for the Treatment of Nasolacrimal Duct Obstruction
Acronym: SLINDO
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: One PI has left University of Michigan; no active work is happening at this time, but when another PI who is well suited is available, the study will resume recruitment.
Sponsor: Thomas Gardner (Other)
Responsible Party: Sponsor-Investigator, Thomas Gardner, Professor of Ophthalmology and Visual Science and Molecular and Integrative Physiology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00114919
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Epiphora; Dacryocystorhinostomy
MeSH Terms: conditions — Lacrimal Apparatus Diseases | interventions — Dacryocystorhinostomy; Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Slit Stent II (Experimental): The Slit Stent II (investigational) device is created by modifying an existing FDA cleared lacrimal stent (BIKA, manufactured by FCI Opthalmics) by adding additional 3 mm and 35 mm long slits of equal depth.
  Interventions: Device: Slit Stent II
- BIKA for DCR (Active Comparator): The BIKA for DCR is a sterile, single-use device, and is an FDA cleared device.
  Interventions: Device: BIKA for DCR

INTERVENTIONS:
Device: Slit Stent II — The Slit-Stent II device is created by modifying the BIKA for DCR lacrimal stent through the addition of a center slit, 12 ± 1.5 mm in length, and two lateral slits 32 ± 4.5 mm in length, each having identical depth measurements to facilitate the drainage of tears. The BIKA for DCR is a sterile, single-use device that is FDA cleared as part of the BIKA family of devices under K911109..There are no changes to the raw materials used in making the modifications to the BIKA for DCR during the manufacturing of the Slit Stent II.
  Other Names: Lacrimal Stent
  Arms: Slit Stent II
Device: BIKA for DCR — The BIKA for DCR lacrimal stent is a bicanalicular intubation device used for intubation of the lacrimal drainage apparatus, especially in cases of dacryocystorhinostomy (conventional or laser). The silicone tube acts as a conformer during the healing process while facilitating drainage of tears through capillary action around the stent. In cases of canalicular lacerations, the silicone tube guides wound healing and prevents the onset of synechia. The BIKA for DCR is a sterile, single-use device, and is an FDA cleared device
  Other Names: stent
  Arms: BIKA for DCR

SUMMARY:
This project aims to test whether a newly designed lacrimal stent - the SlitStent - when placed into the lacrimal system in the standard fashion following a DCR surgery, will provide good symptomatic relief for epiphora and be well tolerated.

Epiphora, or severe tearing, is both a very common debilitating symptom and a potential cause of dangerous infections (i.e. dacryocystitis and orbital cellulitis). DCR+lacrimal stenting surgery is 80-95% successful at improving epiphora, and the longer the stent remains in place, the better the long-term outcome. However, lacrimal stents that provide adequate circumferential force to facilitate post-DCR healing also occupy space and prevent good tear drainage until removed. Yet patients want complete symptomatic improvement as soon as possible, even if it compromises long-term results.

This study aims to test a newly designed lacrimal stent that allows tears to drain through the lumen of the stent. The new stent is constructed by modifying a commercially available stent by placing openings along the side of the stent using a process developed by a University of Michigan engineer/collaborator. Following slit placement, the stent will be gas-sterilized for surgery. Patient who are scheduled for DCR+stenting surgery who provide informed consent will be randomized 2:1 to receive the investigational SlitStent or the standard commercially available stent. Following surgery, patients will be assessed both clinically, which is standard of care, and via a patient questionnaire.

DETAILED DESCRIPTION:
This is a single center study that will be conducted at the University of Michigan (Ann Arbor, Michigan). Fifty (50) subjects will be enrolled and treated with either the experimental Slit Stent II or the control stent BIKA for DCR. Patients who are currently scheduled to undergo a DCR (dacryocystorhinostomy) as per standard of care will be offered participation in the study. Patients who elect to participate in the study will be consented and then randomized to the treatment or control arm.

A lacrimal stent is hollow silicone tubing with a non-traumatic tip. The tubing is securely attached into malleable stainless steel probes that are used to guide the silicone tubing through the lacrimal drainage apparatus. The device is used to maintain an open lacrimal path between the surface of the eye and the nasal passages, particularly during a healing process following injury or surgery.

The BIKA for DCR lacrimal stent is a bicanalicular intubation device used for intubation of the lacrimal drainage apparatus, especially in cases of dacryocystorhinostomy (conventional or laser). The silicone tube acts as a conformer during the healing process while facilitating drainage of tears through capillary action around the stent. In cases of canalicular lacerations, the silicone tube guides wound healing and prevents the onset of synechia.

The BIKA lacrimal stent consists of a single unit including a silicone tube (length: 280 mm, external diameter: 0.94 mm), and one steel probe at each end of the silicone tube (length: 53 mm, external diameter: 0.8 mm) with round tips.

The BIKA for DCR is a sterile, single-use device, and is an FDA cleared device.

The Slit Stent II (investigational) device is created by modifying an existing FDA cleared lacrimal stent (Bika, manufactured by FCI Opthalmics) by adding additional 3 mm and 35 mm long slits of equal depth.

The axial cutouts located on the stent allow drainage of tears from the ocular surface to the nasal/oropharynx cavities through the internal lumen of the stent.

All modifications to the stent are inspected under an optical microscope at a magnification of at least 5x to ensure they are free from cutting defects, which could impact the structural integrity of the Slit Stent II. To ensure that the Slit Stent II can withstand the forces experienced during implantation and removal, additional mechanical integrity tests were performed. Comparing the implantation forces to the maximum insertion and removal force, it was determined that the modified Slit Stent II will have excellent tensile strength - essentially identical to unmodified stent - to prevent mechanical failure in patient use. Each section was tested to determine the maximum elongation and force it can withstand before failure.

The study duration will be 6 months for all study patients.

The following examination schedule will be followed from screening through the postoperative visits:

* Screening (Day -60 to Day 0 Preoperatively)
* Device implantation operation
* Phone call Assessment at 1 day post op
* Phone call Assessment at 45 days post op (+/- 15 days)
* Day 5-14 postoperatively
* Day 30-120 postoperatively (with stent removal)
* 4-7 month final post-operative exam

Subjects will be randomly assigned to the experimental vs. control stents using a randomized block design with 1:1 allocation to treatment and control. Stents will be provided to the surgical team on the day of surgery by the Study Coordinator. Surgical team, recruitment staff, and scheduling staff will be masked to treatment assignment until day of surgery. All tests and measurements should be obtained in accordance with the procedures specified in this protocol. If it is not possible to perform a measurement or examination due to the individual eye's specific ocular pathology, the reason for not performing the test or measurement should be documented on the source documents.

The investigator may designate one or more surgeon sub-investigators at his/her investigative site. A surgeon sub-investigator may evaluate subjects for the study and perform the Slit Stent II lacrimal stent intubation. Surgeon sub-investigators will be listed on all applicable investigator regulatory documents (including the delegation of responsibilities log) and will complete all sponsor-required training for the study.

For the two post-op study visits, the Quality of Life (QOL) questionnaire (Glasgow Benefit Inventory (GBI)- see Appendix A) and the Patient Tearing Questionnaire (Munk Scale and Lac-Q questionnaire, see Appendix B) will be administered by an interviewer, and the interviewer will record the subject's responses directly onto the corresponding questionnaire CRFs or source documents and calculate the GBI score, Munk Score, and Lac-Q score.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to comply with schedule for follow-up visits and postoperative evaluations.
2. Eligible for unilateral DCR surgery with stenting for treatment of epiphora secondary to nasolacrimal duct obstruction.Ability to instill post-operative eye drop
3. Signed written, informed consent.

Exclusion Criteria:

1. Subjects under legal guardianship or who, in the investigator's opinion, lack the mental capacity to provide written informed consent for study participation.
2. Subjects scheduled for bilateral DCR surgery
3. Subjects with known sensitivity to silicone
4. Subjects with a current condition that, in the investigator's opinion, would interfere with the treatment.
5. Inability to use eye drops
6. Subjects with a known sensitivity to required study medications (e.g. antibiotic drops) if an alternative medication is not available.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety, as measured by number of subjects with at least one Adverse Event | Surgery to final exit visit (Month 4-7)
  Adverse events will be recorded from the time of surgical implantation of the device until the final visit. Ophthalmic complications or adverse events that are observed by the investigator or reported by the subject will be recorded on the CRFs. For all adverse effects, sufficient information will be pursued and/or obtained so as to permit 1) an adequate determination of the outcome of the effect (i.e., whether the effect should be classified as a serious adverse effect) and; 2) an assessment of the causal relationship between the adverse effect and the investigational device or, if applicable, the other study treatment or diagnostic product(s).

SECONDARY OUTCOMES:
Glasgow Benefit Inventory (GBI) Questionnaire (Quality of Life) | 1-4 month post-operative follow-up visit
  The effectiveness parameter evaluated will be the mean composite score for the GBI administered post-treatment at the 1-4 month post-operative follow-up visit. scores can range from -100 to 100 where -100 represents decline in symptoms or function and 100 represents greatest improvement.
Lac-Q score | 1-4 months post operative
  The Lac-Q questionnaire, published in 2011, is a patient symptom questionnaire developed for lacrimal drainage surgery.1-2 The questionnaire contains two scores, one is specific for eye-symptoms, and the other assesses the social impact of symptoms. The scores are combined for a single Lac-Q score, whose lowest possible score can be 0 and highest 23, where 0 represents no problems related to watery eyes and 23 represents most symptoms and social challenge from them.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gardner, MD, MS, Principal Investigator — University of Michigan Kellogg Eye Center
Locations (1):
- Kellogg Eye Center, 1000 Wall Street, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No